CLINICAL TRIAL: NCT02402647
Title: Cognitive Rehabilitation and Exposure Therapy for Veterans With Hoarding Disorder
Brief Title: Cognitive Rehab and Exposure Treatment for Hoarding
Acronym: CREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLNA-005-14S
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Hoarding Disorder
Keywords: Hoarding; Compulsive Hoarding
MeSH Terms: conditions — Hoarding Disorder; Hoarding | interventions — Cognitive Training; Implosive Therapy

STUDY DESIGN:
Intervention Model Description: Cognitive rehabilitation and exposure/sorting therapy (CREST) versus Exposure therapy only
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Rehabilitation and Exposure/Sorting Treatment (CREST) (Experimental): Compensatory Cognitive Training (CCT) is a manualized, low-tech, cognitive training intervention designed to target cognitive impairments common in people with psychiatric illness. The CCT modules specifically selected for CREST map onto known areas of HD neurocognitive deficits or weakness and include training in prospective memory, prioritizing, problem solving, planning, and cognitive flexibility.
  Symptoms of acquiring and saving are themselves avoidance behaviors that are performed to avoid internal distress related to negative thoughts and emotions. Avoidance serves to reduce distress related to the beliefs regarding the necessity and utility of possessions. In the CREST condition, the second part and the majority of treatment is dedicated to exposure therapy (ET) for discarding and not acquiring while in the control condition, the entire treatment will consist of ET.
  Interventions: Behavioral: Cognitive Rehabilitation and Exposure/Sorting Treatment (CREST)
- Exposure Therapy (ET) (Active Comparator): The investigators propose to use a robust control condition, exposure therapy (ET), with the same frequency and amount of therapist contact as CREST. Twenty-six weekly, individual ET sessions (6 months) will be delivered. The control group will receive ET for all 26 sessions and no cognitive training. As in CREST, the ET sessions will be manualized and copies utilized during session by both the patient and therapist.
  Interventions: Behavioral: Exposure Therapy (ET)

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation and Exposure/Sorting Treatment (CREST) — Compensatory Cognitive Training is a manualized, low-tech, cognitive training intervention designed to target cognitive impairments common in people with psychiatric illness. The CCT modules specifically selected for CREST map onto known areas of HD neurocognitive deficits or weakness and include training in prospective memory, prioritizing, problem solving, planning, and cognitive flexibility.
  Symptoms of acquiring and saving are themselves avoidance behaviors that are performed to avoid internal distress related to negative thoughts and emotions. Avoidance serves to reduce distress related to the beliefs regarding the necessity and utility of possessions. In the CREST condition, the second part and the majority of treatment is dedicated to exposure therapy (ET) for discarding and not acquiring while in the control condition, the entire treatment will consist of ET.
  Arms: Cognitive Rehabilitation and Exposure/Sorting Treatment (CREST)
Behavioral: Exposure Therapy (ET) — The investigators propose to use a robust control condition, ET, with the same frequency and amount of therapist contact as CREST. Twenty-six weekly, individual ET sessions (6 months) will be delivered. The control group will receive ET for all 26 sessions and no cognitive training. As in CREST, the ET sessions will be manualized and copies utilized during session by both the patient and therapist.
  Arms: Exposure Therapy (ET)

SUMMARY:
This project will utilize a novel behavioral intervention for hoarding disorder that takes into account age and neurocognitive factors. The goal of this project is to gain knowledge on how treatment components may or may not work for Veterans with hoarding disorder. Further, the investigators hope to increase understanding of functional and long term outcomes in response to hoarding treatment.

DETAILED DESCRIPTION:
Objective: The investigators propose to conduct a randomized controlled trial comparing six months (26 sessions) of Cognitive Rehabilitation and Exposure/Sorting Therapy (CREST) treatment to a robust comparator, six months of Exposure Therapy alone, in 136 participants with HD.

Research Design: Assessments will be administered at baseline, during treatment (sessions 7, 13, 21), post-treatment, and 3- and 6-month follow-up, thus, all participants will be enrolled for one year.

Methodology: The primary objective is to evaluate whether CREST significantly reduces hoarding symptoms and improves functional capacity and quality of life when compared to exposure therapy alone. The investigators will also examine the impact of treatment mediators; treatment adherence, changes in executive functioning, avoidance, symptom severity on outcomes. Age and executive functioning will also be explored as potential moderators. Finally, by repeatedly measuring treatment targets, the investigators will examine time to maximum treatment effect in an effort to understand mechanisms of change.

Clinical Relationships: By providing a treatment for many Veterans with HD, the investigators can alter the course of their symptom trajectory and negative consequences, resulting in both healthcare costs savings and improved quality of life for Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Veterans age 18-85
* Hoarding Disorder diagnosis outlined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)6 as measured by the Structured Interview for Hoarding Disorder (SIHD)67
* HD as a primary diagnosis
* Stable on medications for at least 12 weeks, with no pharmacologic changes expected or made during the 12-month study
* Voluntary consent to participate

Exclusion Criteria:

* Diagnosis of:

  * psychotic disorder
  * substance abuse disorder as measured by the Mini-International Neuropsychiatric Interview (M.I.N.I.)68
* Current or history of any neurodegenerative disease
* Active suicidal ideation
* Concurrent participation in psychotherapy or ET for HD, or prior history of CREST for HD

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine R Ayers, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CREST: Compensatory Cognitive Training (CCT) is a manualized, low-tech, cognitive training intervention designed to target cognitive impairments common in people with psychiatric illness. The CCT modules specifically selected for CREST map onto known areas of HD neurocognitive deficits or weakness and include training in prospective memory, prioritizing, problem solving, planning, and cognitive flexibility.
  Symptoms of acquiring and saving are themselves avoidance behaviors that are performed to avoid internal distress related to negative thoughts and emotions. Avoidance serves to reduce distress related to the beliefs regarding the necessity and utility of possessions. In the CREST condition, the second part and the majority of treatment is dedicated to exposure therapy (ET) for discarding and not acquiring while in the control condition, the entire treatment will consist of ET.
- Exposure Therapy: The investigators propose to use a robust control condition, ET, with the same frequency and amount of therapist contact as CREST. Twenty-six weekly, individual ET sessions (6 months) will be delivered. The control group will receive ET for all 26 sessions and no cognitive training. As in CREST, the ET sessions will be manualized and copies utilized during session by both the patient and therapist.
  ET: The investigators propose to use a robust control condition, ET, with the same frequency and amount of therapist contact as CREST. Twenty-six weekly, individual ET sessions (6 months) will be delivered. The control group will receive ET for all 26 sessions and no cognitive training. As in CREST, the ET sessions will be manualized and copies utilized during session by both the patient and therapist.
Period: Overall Study
Arm/Group | CREST | Exposure Therapy
Started | 59 | 56
Completed | 34 | 42
Not Completed | 25 | 14
Not completed — Lost to Follow-up | 13 | 7
Not completed — Protocol Violation | 1 | 1
Not completed — scheduled and timed out | 2 | 1
Not completed — medical illness | 2 | 4
Not completed — Moved | 2 | 0
Not completed — loved one illness | 1 | 0
Not completed — deceased preexisting condition | 2 | 0
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- CREST: CREST: Compensatory Cognitive Training is a manualized, low-tech, cognitive training intervention designed to target cognitive impairments common in people with psychiatric illness. The CCT modules specifically selected for CREST map onto known areas of HD neurocognitive deficits or weakness and include training in prospective memory, prioritizing, problem solving, planning, and cognitive flexibility.
  Symptoms of acquiring and saving are themselves avoidance behaviors that are performed to avoid internal distress related to negative thoughts and emotions. Avoidance serves to reduce distress related to the beliefs regarding the necessity and utility of possessions. In the CREST condition, the second part and the majority of treatment is dedicated to exposure therapy (ET) for discarding and not acquiring while in the control condition, the entire treatment will consist of ET.
- Total: Total of all reporting groups
Arm/Group | CREST | Exposure Therapy | Total
Number analyzed (Participants) | 59 | 56 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (9.1) | 62.8 (12.7) | 61.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 16 | 42
  Male | 33 | 40 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
  Black or African American | 8 | 6 | 14
  White | 37 | 35 | 72
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 5 | 1 | 6
Saving Inventory [Mean (Standard Deviation); unit: units on a scale] — Scores on the SI-R range from 0-92 with a higher score meaning worse hoarding severity
  units on a scale | 59.9 (15.8) | 55.3 (14.8) | 57.7 (15.4)

OUTCOME MEASURES:

1. Primary Outcome: Saving Inventory Revised
Description: Hoarding symptom severity (primary outcome) will be measured using the Savings Inventory-Revised (SI-R)56, a 23-item self-report measure used to assess common hoarding symptoms. Subscales include clutter, acquisition, and difficulty discarding. The SI-R has demonstrated good internal consistency, divergent validity, concurrent validity, and test-retest reliability in clinical samples with hoarding. The total score will be used for analyses. Total of 23 items divided into 3 subscales, each item Likert scale ranges from 0-4 (0= not at all, 4= extreme), Clutter Subscale (9 items): scores greater than 13 indicate clinical significance (Max score=36), Difficulty Discarding/Saving Subscale (7 items): scores greater than 13 indicate clinical significance, Acquisition Subscale (7 items): scores greater than 15 indicate clinical significance (Max Score= 28). Total Max score = 92. A Total score greater than 40 is a typical score for people experiencing challenges with hoarding behaviors.
Time Frame: Baseline to 6 month-follow-up (12 months total)
Population: For SI-R for individual missing responses replace with mean; individuals who missed more than 1/3 of the survey are excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CREST | Exposure Therapy
Number analyzed (Participants) | 59 | 56
score on a scale
  Baseline SI-R:: number analyzed (Participants) | 59 | 55
  Baseline SI-R: | 59.9 (15.8) | 55.3 (14.8)
  Baseline SI-R: Clutter Subcategory | 25.2 (7.7) | 23.0 (8.2)
  Baseline SI-R: Acquisition Subcategory | 16.6 (5.5) | 14.4 (5.4)
  Baseline SI-R: Discarding Subcategory | 18.1 (5.5) | 17.9 (5.1)
  Timepoint 1 (S7) SI-R: number analyzed (Participants) | 48 | 45
  Timepoint 1 (S7) SI-R | 51.6 (16.8) | 50.5 (16.4)
  Timepoint 1 (S7) SI-R: Clutter Subcategory: number analyzed (Participants) | 48 | 45
  Timepoint 1 (S7) SI-R: Clutter Subcategory | 22.6 (8.4) | 21.7 (8.0)
  Timepoint 1 (S7) SI-R: Acquisition Subcategory: number analyzed (Participants) | 48 | 45
  Timepoint 1 (S7) SI-R: Acquisition Subcategory | 14.1 (5.8) | 12.9 (6.1)
  Timepoint 1 (S7) SI-R: Discarding Subcategory: number analyzed (Participants) | 48 | 45
  Timepoint 1 (S7) SI-R: Discarding Subcategory | 14.9 (5.2) | 15.9 (5.0)
  Timepoint 2 (S13) SI-R:: number analyzed (Participants) | 35 | 41
  Timepoint 2 (S13) SI-R: | 47.3 (17.7) | 45.5 (16.9)
  Timepoint 2 (S13) SI-R: Clutter Subcategory: number analyzed (Participants) | 35 | 41
  Timepoint 2 (S13) SI-R: Clutter Subcategory | 20.1 (8.7) | 19.6 (8.5)
  Timepoint 2 (S13) SI-R: Acquisition Subcategory: number analyzed (Participants) | 35 | 41
  Timepoint 2 (S13) SI-R: Acquisition Subcategory | 13.1 (6.3) | 11.5 (6.0)
  Timepoint 2 (S13) SI-R: Discarding Subcategory: number analyzed (Participants) | 35 | 41
  Timepoint 2 (S13) SI-R: Discarding Subcategory | 14.2 (5.5) | 14.4 (5.1)
  Timepoint 3 (S21) SI-R:: number analyzed (Participants) | 29 | 32
  Timepoint 3 (S21) SI-R: | 45.0 (18.9) | 41.1 (17.3)
  Timepoint 3 (S21) SI-R: Clutter Subcategory: number analyzed (Participants) | 29 | 32
  Timepoint 3 (S21) SI-R: Clutter Subcategory | 19.8 (8.3) | 18.1 (7.6)
  Timepoint 3 (S21) SI-R: Acquisition Subcategory: number analyzed (Participants) | 29 | 56
  Timepoint 3 (S21) SI-R: Acquisition Subcategory | 11.7 (6.2) | 9.3 (5.7)
  Timepoint 3 (S21) SI-R: Discarding Subcategory: number analyzed (Participants) | 29 | 32
  Timepoint 3 (S21) SI-R: Discarding Subcategory | 13.5 (7.0) | 13.8 (5.7)
  Post-Treatment SI-R:: number analyzed (Participants) | 29 | 37
  Post-Treatment SI-R: | 37 (19.6) | 29.9 (18.6)
  Post-Treatment SI-R: Clutter Subcategory: number analyzed (Participants) | 29 | 37
  Post-Treatment SI-R: Clutter Subcategory | 16.1 (9.4) | 12.9 (8.8)
  Post-Treatment SI-R: Acquisition Subcategory: number analyzed (Participants) | 29 | 37
  Post-Treatment SI-R: Acquisition Subcategory | 10.0 (6.1) | 7.3 (5.9)
  Post-Treatment SI-R: Discarding Subcategory: number analyzed (Participants) | 29 | 37
  Post-Treatment SI-R: Discarding Subcategory | 10.9 (6.4) | 9.8 (5.8)
  3 month post-treatment SI-R:: number analyzed (Participants) | 21 | 28
  3 month post-treatment SI-R: | 37.5 (21.4) | 32.6 (20.4)
  3 month post-treatment SI-R: Clutter Subcategory: number analyzed (Participants) | 21 | 28
  3 month post-treatment SI-R: Clutter Subcategory | 16.2 (10.5) | 14.5 (8.9)
  3 month post-treatment SI-R: Acquisition Subcategory: number analyzed (Participants) | 21 | 28
  3 month post-treatment SI-R: Acquisition Subcategory | 9.9 (6.5) | 7.9 (6.3)
  3 month post-treatment SI-R: Discarding Subcategory: number analyzed (Participants) | 21 | 28
  3 month post-treatment SI-R: Discarding Subcategory | 11.3 (7.3) | 10.2 (6.4)
  6 month post-treatment SI-R:: number analyzed (Participants) | 22 | 29
  6 month post-treatment SI-R: | 34.3 (18.1) | 28.9 (18.9)
  6 month post-treatment SI-R: Clutter Subcategory: number analyzed (Participants) | 22 | 29
  6 month post-treatment SI-R: Clutter Subcategory | 15.2 (9.3) | 12.2 (9.0)
  6 month post-treatment SI-R: Acquisition Subcategory: number analyzed (Participants) | 22 | 29
  6 month post-treatment SI-R: Acquisition Subcategory | 8.7 (5.2) | 6.7 (5.7)
  6 month post-treatment SI-R: Discarding Subcategory: number analyzed (Participants) | 22 | 29
  6 month post-treatment SI-R: Discarding Subcategory | 10.3 (6.7) | 9.9 (5.8)

2. Secondary Outcome: UCSD Performance-Based Skills Assessment (UPSA)
Description: The University of California San Diego (UCSD) Performance-Based Skills Assessment (UPSA)76 is an assessment of everyday functioning skills including household skills (e.g., writing a shopping list based on a recipe, range 0 to 4), communication (e.g., rescheduling appointments, range 0 to 12), finance (e.g., paying a utility bill, range 0 to 11), comprehension and planning (e.g., planning outings, range 0 to 14), and transportation (e.g., comprehension of a bus schedule, range 0 to 9). The subscales are scored, converted to a percentage, and weighed equally toward the total score of 100; higher score equals better performance for all subscales and total. The UPSA has demonstrated high inter-rater reliability (0.91) and convergent validity with other performance-based measures. The total UPSA summary score will be used for analyses. *Nearly half of each timepoint was out of 60 due to adjustments for COVID-19, a total of 60 was used with financial, communication, and planning subscales.
Time Frame: Baseline to 6 months post-treatment (on average 1 year)
Population: As the study progressed participants may have dropped out/left or refused to complete/answer and questions/tasks associated
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CREST | Exposure Therapy
Number analyzed (Participants) | 59 | 56
score on a scale
  Baseline UPSA: number analyzed (Participants) | 58 | 56
  Baseline UPSA | 49.0 (7.4) | 49.1 (6.8)
  Baseline UPSA: Financial Subcategory: number analyzed (Participants) | 58 | 56
  Baseline UPSA: Financial Subcategory | 18.3 (2.5) | 18.0 (2.2)
  Baseline UPSA: Communication Subcategory: number analyzed (Participants) | 58 | 56
  Baseline UPSA: Communication Subcategory | 16.2 (2.6) | 15.3 (3.1)
  Baseline UPSA: Comprehension/Planning Subcategory: number analyzed (Participants) | 58 | 56
  Baseline UPSA: Comprehension/Planning Subcategory | 14.5 (5.2) | 15.8 (4.2)
  Baseline UPSA: Transportation Subcategory: number analyzed (Participants) | 47 | 47
  Baseline UPSA: Transportation Subcategory | 16.2 (2.8) | 15.9 (3.8)
  Baseline UPSA: Household Skills Subcategory: number analyzed (Participants) | 47 | 47
  Baseline UPSA: Household Skills Subcategory | 17.6 (3.7) | 18.5 (2.3)
  Timepoint 1 (S7) UPSA: number analyzed (Participants) | 43 | 41
  Timepoint 1 (S7) UPSA | 50.3 (8.3) | 50.9 (6.4)
  Timepoint 1 (S7) UPSA: Financial Subcategory: number analyzed (Participants) | 41 | 41
  Timepoint 1 (S7) UPSA: Financial Subcategory | 18.8 (1.5) | 18.3 (2.3)
  Timepoint 1 (S7) UPSA: Communication Subcategory: number analyzed (Participants) | 43 | 41
  Timepoint 1 (S7) UPSA: Communication Subcategory | 15.9 (3.0) | 16.6 (2.0)
  Timepoint 1 (S7) UPSA: Comprehension/Planning Subcategory: number analyzed (Participants) | 43 | 41
  Timepoint 1 (S7) UPSA: Comprehension/Planning Subcategory | 16.4 (3.5) | 16.0 (4.6)
  Timepoint 1 (S7) UPSA: Transportation Subcategory: number analyzed (Participants) | 33 | 34
  Timepoint 1 (S7) UPSA: Transportation Subcategory | 15.9 (2.7) | 16.6 (2.9)
  Timepoint 1 (S7) UPSA: Household Skills Subcategory: number analyzed (Participants) | 33 | 33
  Timepoint 1 (S7) UPSA: Household Skills Subcategory | 18.3 (2.7) | 18.0 (2.8)
  Timepoint 2 (S13) UPSA: number analyzed (Participants) | 30 | 35
  Timepoint 2 (S13) UPSA | 52.7 (4.0) | 52.7 (5.2)
  Timepoint 2 (S13) UPSA: Financial Subcategory: number analyzed (Participants) | 30 | 35
  Timepoint 2 (S13) UPSA: Financial Subcategory | 18.6 (1.7) | 1.1 (2.5)
  Timepoint 2 (S13) UPSA: Communication Subcategory: number analyzed (Participants) | 30 | 35
  Timepoint 2 (S13) UPSA: Communication Subcategory | 16.7 (2.4) | 16.8 (2.4)
  Timepoint 2 (S13) UPSA: Comprehension/Planning Subcategory: number analyzed (Participants) | 30 | 35
  Timepoint 2 (S13) UPSA: Comprehension/Planning Subcategory | 17.4 (3.2) | 17.8 (3.2)
  Timepoint 2 (S13) UPSA: Transportation Subcategory: number analyzed (Participants) | 22 | 29
  Timepoint 2 (S13) UPSA: Transportation Subcategory | 16.0 (2.5) | 16.8 (2.6)
  Timepoint 2 (S13) UPSA: Household Skills Subcategory: number analyzed (Participants) | 22 | 29
  Timepoint 2 (S13) UPSA: Household Skills Subcategory | 17.1 (4.0) | 17.6 (2.9)
  Timepoint 3 (S21) UPSA: number analyzed (Participants) | 30 | 35
  Timepoint 3 (S21) UPSA | 52.7 (4.0) | 52.7 (5.2)
  Timepoint 3 (S21) UPSA: Financial Subcategory: number analyzed (Participants) | 30 | 35
  Timepoint 3 (S21) UPSA: Financial Subcategory | 18.6 (1.7) | 18.1 (2.5)
  Timepoint 3 (S21) UPSA: Communication Subcategory: number analyzed (Participants) | 30 | 35
  Timepoint 3 (S21) UPSA: Communication Subcategory | 16.7 (2.4) | 16.8 (2.4)
  Timepoint 3 (S21) UPSA: Comprehension/Planning Subcategory: number analyzed (Participants) | 30 | 35
  Timepoint 3 (S21) UPSA: Comprehension/Planning Subcategory | 17.4 (3.2) | 17.8 (3.2)
  Timepoint 3 (S21) UPSA: Transportation Subcategory: number analyzed (Participants) | 22 | 29
  Timepoint 3 (S21) UPSA: Transportation Subcategory | 16.0 (2.5) | 16.8 (2.6)
  Timepoint 3 (S21) UPSA: Household Skills Subcategory: number analyzed (Participants) | 22 | 29
  Timepoint 3 (S21) UPSA: Household Skills Subcategory | 17.1 (4.0) | 17.6 (2.9)
  Post Treatment UPSA: number analyzed (Participants) | 22 | 27
  Post Treatment UPSA | 51.8 (7.2) | 54.6 (5.2)
  Post Treatment UPSA: Financial Subcategory: number analyzed (Participants) | 22 | 27
  Post Treatment UPSA: Financial Subcategory | 18.3 (2.4) | 18.9 (1.7)
  Post Treatment UPSA: Communication Subcategory: number analyzed (Participants) | 22 | 27
  Post Treatment UPSA: Communication Subcategory | 16.3 (3.0) | 17.8 (1.7)
  Post Treatment UPSA: Comprehension/Planning Subcategory: number analyzed (Participants) | 22 | 27
  Post Treatment UPSA: Comprehension/Planning Subcategory | 17.2 (4.6) | 17.9 (3.4)
  Post Treatment UPSA: Transportation Subcategory: number analyzed (Participants) | 15 | 21
  Post Treatment UPSA: Transportation Subcategory | 16.8 (2.1) | 17.0 (2.4)
  Post Treatment UPSA: Household Skills Subcategory: number analyzed (Participants) | 15 | 21
  Post Treatment UPSA: Household Skills Subcategory | 17.3 (4.2) | 18.3 (2.4)
  3 month Follow Up UPSA: number analyzed (Participants) | 11 | 22
  3 month Follow Up UPSA | 54.1 (4.5) | 54.0 (3.3)
  3 month Follow Up UPSA: Financial Subcategory: number analyzed (Participants) | 11 | 22
  3 month Follow Up UPSA: Financial Subcategory | 18.6 (2.1) | 18.8 (1.3)
  3 month Follow Up UPSA: Communication Subcategory: number analyzed (Participants) | 11 | 22
  3 month Follow Up UPSA: Communication Subcategory | 16.6 (2.7) | 17.2 (1.8)
  3 month Follow Up UPSA: Comprehension/Planning Subcategory: number analyzed (Participants) | 11 | 22
  3 month Follow Up UPSA: Comprehension/Planning Subcategory | 18.9 (1.9) | 18.7 (2.6)
  3 month Follow Up UPSA: Transportation Subcategory: number analyzed (Participants) | 8 | 19
  3 month Follow Up UPSA: Transportation Subcategory | 15.2 (6.5) | 17.4 (2.7)
  3 month Follow Up UPSA: Household Skills Subcategory: number analyzed (Participants) | 8 | 19
  3 month Follow Up UPSA: Household Skills Subcategory | 15.6 (6.8) | 16.6 (5.3)
  6 month Follow Up UPSA:: number analyzed (Participants) | 11 | 20
  6 month Follow Up UPSA: | 52.5 (7.4) | 53.8 (5.0)
  6 month Follow Up UPSA: Financial Subcategory: number analyzed (Participants) | 11 | 20
  6 month Follow Up UPSA: Financial Subcategory | 19.1 (1.4) | 18.9 (1.4)
  6 month Follow Up UPSA: Communication Subcategory: number analyzed (Participants) | 11 | 20
  6 month Follow Up UPSA: Communication Subcategory | 15.8 (4.1) | 17.3 (2.7)
  6 month Follow Up UPSA: Comprehension/Planning Subcategory: number analyzed (Participants) | 11 | 20
  6 month Follow Up UPSA: Comprehension/Planning Subcategory | 17.5 (4.3) | 17.6 (3.0)
  6 month Follow Up UPSA: Transportation Subcategory: number analyzed (Participants) | 7 | 19
  6 month Follow Up UPSA: Transportation Subcategory | 14.0 (6.5) | 18.0 (2.3)
  6 month Follow Up UPSA: Household Skills Subcategory: number analyzed (Participants) | 7 | 19
  6 month Follow Up UPSA: Household Skills Subcategory | 20.0 (0.0) | 17.6 (3.1)

3. Secondary Outcome: UCSD SORT Test
Description: The UCSD SORT Test (U-SORT) is a cognitive test that will be used to measure Veteran participants' organizational skills as they relate to functional capacity. During the administration of the U-SORT, participants are instructed to sort 42 household objects (e.g., bent and unbent paper clips, used and unused condiment packets) from a hypothetical "junk drawer" into either "keep" or "trash" piles. Each item has a correct response and participants are given two minutes to complete the task and one point is awarded for each correctly sorted item, for a total of 42 points (range of 0 to 42). A higher total score indicates a higher level of organizational skills. The U-SORT has high internal consistency (? = .86) and adequate convergent validity. The total U-SORT score will be used in analyses.
Time Frame: Baseline to 6 months post-treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cognitive Rehabilitation and Exposure/Sorting Therapy: Compensatory Cognitive Training (CCT) is a manualized, low-tech, cognitive training intervention designed to target cognitive impairments common in people with psychiatric illness. The CCT modules specifically selected for CREST map onto known areas of HD neurocognitive deficits or weakness and include training in prospective memory, prioritizing, problem solving, planning, and cognitive flexibility.
  Symptoms of acquiring and saving are themselves avoidance behaviors that are performed to avoid internal distress related to negative thoughts and emotions. In the CREST condition, the second part and the majority of treatment is dedicated to exposure therapy (ET) for discarding and not acquiring while in the control condition, the entire treatment will consist of ET.
- Exposure Therapy: Exposure Therapy: The investigators propose to use a robust control condition, ET, with the same frequency and amount of therapist contact as CREST. Twenty-six weekly, individual ET sessions (6 months) will be delivered. The control group will receive ET for all 26 sessions and no cognitive training. As in CREST, the ET sessions will be manualized and copies utilized during session by both the patient and therapist.
Arm/Group | Cognitive Rehabilitation and Exposure/Sorting Therapy | Exposure Therapy
Number analyzed (Participants) | 59 | 56
score on a scale
  Baseline USORT | 33.1 (3.9) | 31.2 (4.7)
  Timepoint 1 (S7) USORT: number analyzed (Participants) | 44 | 41
  Timepoint 1 (S7) USORT | 32.5 (5.0) | 32.7 (5.3)
  Timepoint 2 (S13) USORT: number analyzed (Participants) | 30 | 35
  Timepoint 2 (S13) USORT | 34.2 (4.1) | 34.2 (4.2)
  Timepoint 3 (S21) USORT: number analyzed (Participants) | 22 | 24
  Timepoint 3 (S21) USORT | 33.2 (6.1) | 32.9 (4.4)
  Post-Treatment USORT: number analyzed (Participants) | 21 | 27
  Post-Treatment USORT | 34.5 (3.4) | 32.3 (5.2)
  3 month Post-Treatment USORT: number analyzed (Participants) | 11 | 22
  3 month Post-Treatment USORT | 36.1 (4.0) | 31.4 (6.9)
  6 month Post-Treatment USORT: number analyzed (Participants) | 11 | 20
  6 month Post-Treatment USORT | 35.9 (2.9) | 34.0 (5.2)

4. Secondary Outcome: Specific Levels of Functioning Test (SLOF)
Description: Self-reported functioning (secondary outcome) will be assessed with the Specific Levels of Functioning test (SLOF)78, a 43-item Likert scale questionnaire with higher scores indicating higher levels of functioning. Subscales include interpersonal relationships (score range of 7 to 35), social acceptability (score range of 6 to 30), participation in activities (score range of 11 to 55), and work skills (score range of 6 to 30). Total of 30 items across four categories and each item ranges from the scale of 1-5 (higher values= better outcomes). Category A. Interpersonal Relationships (items 1-7): 5= Highly Typical, 1= Highly Untypical. Category B. Social Acceptability (items 8-13): 5= Never, 1= Always. Category C. Activities (items 14-24): 5= Totally Self Sufficient, 1= No Opportunity to perform. Category D. Work Skills (items 25-30): 5= Highly Typical, 1= Highly Untypical. Total Max Score Range= 30-150).The SLOF has demonstrated excellent reliability and internal consistency.
Time Frame: Baseline to 6 months post-treatment
Population: For SLOF regarding individual missing responses replaced with mean; individuals who missed more than 1/3 of the survey are excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Exposure Therapy: The investigators propose to use a robust control condition, Exposure Therapy (ET), with the same frequency and amount of therapist contact as CREST. Twenty-six weekly, individual ET sessions over the course of 6 months will be delivered. The control group will receive ET for all 26 sessions and no cognitive training. As in CREST, the ET sessions will be manualized and copies utilized during session by both the patient and therapist.
Arm/Group | CREST | Exposure Therapy
Number analyzed (Participants) | 59 | 56
score on a scale
  Baseline SLOF Overall | 123.9 (12.9) | 128.0 (15.0)
  Baseline Interpersonal Relationships Subscale | 25.6 (6.2) | 24.7 (7.0)
  Baseline Social Acceptability Subscale | 26.6 (2.5) | 26.7 (2.5)
  Baseline Activities Subscale | 50.7 (4.8) | 51.8 (5.7)
  Baseline Work Skills Subscale: number analyzed (Participants) | 58 | 55
  Baseline Work Skills Subscale | 24.5 (4.9) | 25.2 (4.9)
  Timepoint 1 (S7) SLOF Overall: number analyzed (Participants) | 45 | 45
  Timepoint 1 (S7) SLOF Overall | 127.0 (15.2) | 128.1 (13.9)
  Timepoint 1 (S7) Interpersonal Relationships Subscale: number analyzed (Participants) | 46 | 45
  Timepoint 1 (S7) Interpersonal Relationships Subscale | 23.1 (6.7) | 24.4 (7.0)
  Timepoint 1 (S7) Social Acceptability Subscale: number analyzed (Participants) | 46 | 45
  Timepoint 1 (S7) Social Acceptability Subscale | 26.8 (2.7) | 27.4 (2.0)
  Timepoint 1 (S7) Activities Subscale: number analyzed (Participants) | 46 | 45
  Timepoint 1 (S7) Activities Subscale | 52.1 (4.4) | 52.2 (4.3)
  Timepoint 1 (S7) Work Skills Subscale: number analyzed (Participants) | 46 | 45
  Timepoint 1 (S7) Work Skills Subscale | 25.0 (4.9) | 24.2 (5.2)
  Timepoint 2 (S13) SLOF Overall: number analyzed (Participants) | 34 | 41
  Timepoint 2 (S13) SLOF Overall | 128.5 (14.6) | 126.0 (15.0)
  Timepoint 2 (S13) Interpersonal Relationships Subscale: number analyzed (Participants) | 34 | 41
  Timepoint 2 (S13) Interpersonal Relationships Subscale | 23.8 (6.4) | 23.4 (6.5)
  Timepoint 2 (S13) Social Acceptability Subscale: number analyzed (Participants) | 34 | 41
  Timepoint 2 (S13) Social Acceptability Subscale | 27.5 (2.3) | 27.0 (2.0)
  Timepoint 2 (S13) Activities Subscale: number analyzed (Participants) | 34 | 41
  Timepoint 2 (S13) Activities Subscale | 52.3 (5.2) | 51.9 (5.3)
  Timepoint 2 (S13) Work Skills Subscale: number analyzed (Participants) | 34 | 41
  Timepoint 2 (S13) Work Skills Subscale | 25.0 (4.7) | 23.6 (5.8)
  Timepoint 3 (S21) SLOF Overall: number analyzed (Participants) | 28 | 32
  Timepoint 3 (S21) SLOF Overall | 128.3 (14.5) | 125.4 (14.8)
  Timepoint 3 (S21) Interpersonal Relationships Subscale: number analyzed (Participants) | 28 | 32
  Timepoint 3 (S21) Interpersonal Relationships Subscale | 24.4 (6.7) | 23.7 (6.8)
  Timepoint 3 (S21) Social Acceptability Subscale: number analyzed (Participants) | 28 | 32
  Timepoint 3 (S21) Social Acceptability Subscale | 26.6 (4.6) | 27.2 (2.1)
  Timepoint 3 (S21) Activities Subscale: number analyzed (Participants) | 28 | 32
  Timepoint 3 (S21) Activities Subscale | 51.7 (4.9) | 51.3 (5.2)
  Timepoint 3 (S21) Work Skills Subscale: number analyzed (Participants) | 28 | 32
  Timepoint 3 (S21) Work Skills Subscale | 25.6 (3.8) | 23.3 (5.3)
  Post-Treatment SLOF Overall: number analyzed (Participants) | 27 | 35
  Post-Treatment SLOF Overall | 131.9 (15.4) | 124.6 (15.9)
  Post-Treatment Interpersonal Relationships Subscale: number analyzed (Participants) | 27 | 35
  Post-Treatment Interpersonal Relationships Subscale | 25.3 (7.1) | 23.2 (7.0)
  Post-Treatment Social Acceptability Subscale: number analyzed (Participants) | 27 | 35
  Post-Treatment Social Acceptability Subscale | 28.0 (2.0) | 27.2 (2.3)
  Post-Treatment Activities Subscale: number analyzed (Participants) | 27 | 35
  Post-Treatment Activities Subscale | 51.8 (8.3) | 51.3 (5.3)
  Post-Treatment Work Skills Subscale: number analyzed (Participants) | 27 | 35
  Post-Treatment Work Skills Subscale | 26.8 (3.7) | 22.9 (5.9)
  3 month Follow Up SLOF Overall: number analyzed (Participants) | 19 | 28
  3 month Follow Up SLOF Overall | 133.9 (11.9) | 125.6 (16.8)
  3 month Follow Up Interpersonal Relationships Subscale: number analyzed (Participants) | 19 | 28
  3 month Follow Up Interpersonal Relationships Subscale | 25.6 (7.4) | 23.8 (6.9)
  3 month Follow Up Social Acceptability Subscale: number analyzed (Participants) | 19 | 28
  3 month Follow Up Social Acceptability Subscale | 28.0 (1.8) | 27.1 (2.4)
  3 month Follow Up Activities Subscale: number analyzed (Participants) | 19 | 28
  3 month Follow Up Activities Subscale | 53.7 (3.7) | 51.6 (5.3)
  3 month Follow Up Work Skills Subscale: number analyzed (Participants) | 19 | 28
  3 month Follow Up Work Skills Subscale | 26.6 (3.9) | 23.1 (6.3)
  6 month Follow Up SLOF Overall: number analyzed (Participants) | 20 | 29
  6 month Follow Up SLOF Overall | 133.2 (13.6) | 124.0 (20.0)
  6 month Follow Up Interpersonal Relationships Subscale: number analyzed (Participants) | 20 | 29
  6 month Follow Up Interpersonal Relationships Subscale | 25.8 (7.0) | 24.6 (6.5)
  6 month Follow Up Social Acceptability Subscale: number analyzed (Participants) | 19 | 29
  6 month Follow Up Social Acceptability Subscale | 27.6 (2.2) | 27.7 (1.9)
  6 month Follow Up Activities Subscale: number analyzed (Participants) | 20 | 28
  6 month Follow Up Activities Subscale | 54.4 (1.8) | 50.9 (6.5)
  6 month Follow Up Work Skills Subscale: number analyzed (Participants) | 20 | 28
  6 month Follow Up Work Skills Subscale | 26.8 (4.0) | 23.5 (7.0)

ADVERSE EVENTS:
Time Frame: Baseline assessment throughout intervention completion (approximately 6-months) and throughout follow-up period (another 6 months) for a total of approximately 1 year.
Arm/Group | Cognitive Rehabilitation and Exposure/Sorting Therapy | Exposure Therapy
All-Cause Mortality (participants affected / at risk) | 2/59 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/56
Other Adverse Events (participants affected / at risk) | 0/59 | 0/56

LIMITATIONS AND CAVEATS:
The addition of motivational interviewing techniques prior to study initiation greatly reduced drop outs. Further, the last half of the study employed licensed clinicians. Finally, due to COVID-19, the study was shut down for several months while we transitioned to all virtual care. During that time, we lost participants to follow-up and those who preferred in person care only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT02402647/Prot_SAP_000.pdf